CLINICAL TRIAL: NCT01751334
Title: Comparison of the Tibiofemoral Rotational Alignment After Mobile and Fixed Bearing Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUHOSKNEE01-RPFLPSF
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty; Replacement; Knee; Rotational Alignment
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile Bearing (Experimental): Mobile bearing total knee arthroplasty
  Interventions: Device: total knee arthroplasty
- Fixed Bearing (Active Comparator): Fixed Bearing total knee arthroplasty
  Interventions: Device: total knee arthroplasty

INTERVENTIONS:
Device: total knee arthroplasty — Mobile Bearing Total knee Arthroplasty
  Other Names: Sigma® RP-F Knee System, Depuy J&J, Warsaw, IN, USA
  Arms: Mobile Bearing
Device: total knee arthroplasty — Fixed Total Knee Arthroplasty
  Other Names: Nexgen® Legacy® Knee LPS-Flex, Zimmer, Warsaw, IN, USA
  Arms: Fixed Bearing

SUMMARY:
The anatomic landmark for the anteroposterior (AP) axis of the proximal tibia and its variability was investigated in this study in order to determine whether a certain landmark could be employed as a reference axis for the proximal tibia after rotating platform mobile bearing (RP-MB) and fixed bearing (FB) total knee arthroplasties (TKAs).

DETAILED DESCRIPTION:
Reference of tibial AP axis for implanting tibial component in total knee arthroplasty have not been concluded. This study can suggest appropriate method for alingning the tibial component to accurate tibial AP axis.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis

Exclusion Criteria:

* infection
* inflammatory arthritis
* reoperation
* severe deformity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-09; Primary Completion 2006-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Tibial anteroposterior axis relative to femoral anteroposterior axis | postoperative 2 weeks
  Tibial anteroposterior axis relative to femoral anteroposterior axis on Computed tomogram images

CONTACTS AND LOCATIONS:
Overall Officials: Sahnghoon Lee, M.D., Ph.D., Principal Investigator; Myung Chul Lee, M.D., Ph.D., Study Chair